CLINICAL TRIAL: NCT00334620
Title: Effectiveness of Radon Spa Therapy in Multimodal Rehabilitative Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forschungsinstitut für Balneologie und Kurortwissenschaft Bad Elster (Other Government)
Collaborators: In-patient rehabilition hospital Klinik Bad Brambach (Unknown); University hospital Dresden, III. Medical hospital and Outpatient clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-3I_1998
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2006-06-08 (Estimated); Status verified 2005-11

CONDITIONS: Rheumatoid Arthritis
Keywords: randomised double-blinded trial; rehabilitation; radon spa therapy; long-term effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Procedure: 15 radon(+CO2) baths vs 15 CO2 baths; beside rehabilitation

SUMMARY:
The study aimed to investigate effects of radon (plus CO2) baths on RA in contrast to artificial CO2 baths in RA rehabilitation.

134 patients of an in-patient rehabilitative programme were randomly assigned to the groups. Outcomes were limitations in occupational context/ daily living (main outcome), pain, medication, etc. measured before start, after end of treatment, and up to a year thereafter.

Superiority of radon treatment was found regarding reduced limitations in daily living until 12 months after end of treatment. Steroid consumption and NSAIDs were significantly reduced.

DETAILED DESCRIPTION:
Objective: To replicate former observed beneficial effects of Radon (plus CO2) baths on RA in contrast to artificial CO2 baths and to investigate its long-term effectiveness and impact on drug consumption.

Methods: Randomised double-blinded trial with 2 randomised balanced groups enrolling 134 patients of an in-patient rehabilitative programme (a 3rd non-randomised group of 73 consecutive patients is not reported here). Outcomes were limitations in occupational context/ daily living, pain, functional capacity, morning stiffness and medication measured before start, after end of treatment, and quarterly in the year thereafter. Repeated-measures analysis of covariance (RM-ANCOVA) of intent-to treat population was performed to investigate treatment effects. Hierarchically ordered hypotheses ensured adherence of the nominal significance level and allowed examining of long-term effects. Starting with all measures until 6 months' follow-up, significant main effects for group allocation (GME) or significant group x course-interactions (GxC) were regarded essential to add the next follow-up for analysis.

Results: Radon treatment resulted in significantly lower limitations of daily living over at least 9 months whereas reference patients returned to baseline level after 6 months already (RM-ANCOVA until 6 months: pGME=.15, pGxC=.016/ 9 months: pGME=.11, pGxC=.025/ 12 months: pGME=.17, pGxC=.033). Furthermore, consumption of steroids and NSAID was remarkably reduced in the Radon group (RM-ANCOVA until 12 months: for steroids pGME=.064, interaction pGxC=.025, maximum difference after 12 months; for NSAID pGME=.035, interaction pGxC=.008, maximum difference after 9 months).

Conclusion: Results suggest beneficial long-term effects of Radon baths as adjunct to a multimodal rehabilitative treatment of RA.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to the 1987 revised ACR criteria for RA

Exclusion Criteria:

* current exacerbations of the inflammatory process
* other systemic inflammatory diseases
* concomitant musculo-skeletal diseases possibly interfering with outcome measurement,
* pregnancy or breast feeding
* disorders of the central nervous system
* a known tendency toward thrombosis
* malignant hypertension
* coronary heart disease
* heart failure, arrhythmia
* severe disorders of lungs, kidneys, or liver
* advanced malignancies
* abuse of alcohol or drugs,
* major skin lesions,
* severe fever, or infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 1998-07; Study Completion 2005-05

PRIMARY OUTCOMES:
limitations in everyday life and private activities
limitations in the occupational context (not for pensioners)
(both self-assessed on 2 100mm-VAS, averaged into 1 criterion if applicable)

SECONDARY OUTCOMES:
pain intensity
pain frequency
morning stiffness
functional capacity
drug consumption (steroids; NSAIDs; DMARDs only descriptively)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Egbert Schröder, MD, Prof, Principal Investigator — Director III. Med. Hospital, University hospital, Technical University Dresden,
Locations (1):
- Klinik Bad Brambach, Bad Brambach, Saxony, Germany

REFERENCES:
- [Background] Franke A, Reiner L, Pratzel HG, Franke T, Resch KL. Long-term efficacy of radon spa therapy in rheumatoid arthritis--a randomized, sham-controlled study and follow-up. Rheumatology (Oxford). 2000 Aug;39(8):894-902. doi: 10.1093/rheumatology/39.8.894. PMID 10952746